CLINICAL TRIAL: NCT05814497
Title: Supraspinal Processing of Sensory Aspects of Pain
Acronym: SCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Robert Coghill, Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-0556
Record Dates: First submitted 2023-02-10; First posted 2023-04-18 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-01

CONDITIONS: Migraine in Children; Complex Regional Pain Syndromes; Musculoskeletal Pain; Functional Abdominal Pain Syndrome; Fibromyalgia
Keywords: chronic pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Musculoskeletal Pain; Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy Controls (Experimental): Healthy controls with no history of chronic pain.
  Interventions: Other: Multisensory Task; Other: Graphesthesia; Other: Divided attention
- Headache and Migraine (Experimental): Individuals who have migraine with headaches.
  Interventions: Other: Multisensory Task; Other: Graphesthesia; Other: Divided attention
- Functional Abdominal Pain Disorder (FAPD) (Experimental): Individuals who have functional abdominal pain disorder.
  Interventions: Other: Multisensory Task; Other: Graphesthesia; Other: Divided attention
- Localized and Diffuse/Widespread Musculoskeletal Pain (MSK) (Experimental): Individuals with chronic musculoskeletal pain.
  Interventions: Other: Multisensory Task; Other: Graphesthesia; Other: Divided attention
- Complex Regional Pain Syndrome (CRPS) (Experimental): Individuals with complex regional pain syndrome.
  Interventions: Other: Multisensory Task; Other: Graphesthesia; Other: Divided attention

INTERVENTIONS:
Other: Multisensory Task — Reversing checkerboard, tones, and finger opposition.
Other: Graphesthesia — Trace numbers on skin.
Other: Divided attention — Divide attention between two noxious stimuli.

SUMMARY:
The goal of this basic science study is to learn about the brain mechanisms of chronic pain across different chronic pain syndromes in pediatric patients. The main questions it aims to answer are:

* Are there shared and distinct brain systems engaged by different forms of pediatric chronic pain?
* What are predictors of recovery from chronic pain?
* What brain systems are associated with the spread of pain?

For this study participants will undergo:

* Functional Magnetic Resonance Imaging (fMRI)
* Quantitative Sensory Testing
* Psychological Assessments

DETAILED DESCRIPTION:
Chronic pain affects approximately 20% of both adults and children in the US and is a source of substantial disability and health care costs. Chronic pain can be challenging to diagnose due to the presence of poorly understood symptoms. When diagnosed, current pharmacologic treatments for pain are remarkably ineffective, while effective non-pharmacologic treatments remain under-utilized. These shortcomings in the diagnosis and treatment of pain arise from tremendous gaps in our knowledge about the basic central nervous system systems that process nociceptive information and instantiate an experience of pain. These gaps are further amplified in the case of pediatric chronic pain due to a lack of basic/translational research. The team of basic scientists and clinician scientists is uniquely positioned to perform human pediatric studies integrating functional neuroimaging with quantitative sensory testing and psychological assessments to delineate brain systems engaged during chronic pain. The study will examine four distinct chronic pain syndromes: migraine, complex regional pain syndrome, functional abdominal pain, and musculoskeletal pain. The study seeks to 1) Identify shared and distinct brain systems engaged by different forms of pediatric chronic pain, 2) Determine if predictors of recovery differ across different chronic pain conditions, 3) Delineate brain systems associated with the spread of pain. To accomplish these aims, the study will recruit 400 patients with chronic pain and 100 healthy participants (age range 10-17). The study will follow all participants longitudinally for 1 year after initiation of treatment to assess the degree of recovery and spread of pain. This basic science investigation will provide a critical foundation of basic knowledge for future clinical trials of diagnostic markers for different forms of chronic pain and for the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients will need a diagnosis of a chronic pain derived congruent with ICD-11 criteria related to headache (migraine, daily headache), abdominal (FAPD), localized MSK (single limb/joint, low back or chest pain), diffuse MSK (widespread MSK pain), or CRPS
* If on medications, they need to be on stable doses of prescribed pain and/or psychiatric medications for 4 weeks before the baseline study visit.
* Male or female, age 10 -17 (inclusive)
* English speaking, able to complete interviews and questionnaires in English

Exclusion Criteria:

* Weight/size incompatible with MRI scanner
* Orthodontic braces, metallic or electronic implants, or other metal objects in the body which obscure or interfere with the MRI, or pose a risk from heating, movement, or malfunction in the MRI environment
* Claustrophobia
* Youth who are pregnant
* Any comorbid rheumatic disease, diagnosis of epilepsy, other neurological diseases, or medical condition (e.g. diabetes, cancer, IBD)
* Present psychiatric disease as defined by DSM IV (e.g. psychosis, bipolar disorder, major depression, generalized anxiety disorder), alcohol or drug dependence, or documented developmental delays or impairments (e.g., autism, cerebral palsy, ADHD, or mental retardation) that, in the opinion of the investigator, would interfere with adherence to study requirements or safe participation in the study
* Skin conditions or past skin damage on the arms or legs in or near sites of sensory testing
* Outside the age range (9 years old or younger; 18 years or older) at the time of consent
* History of > 1 month opioid treatment.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
FMRI: BOLD resting connectivity of the amygdala | Baseline
  BOLD resting connectivity of the amygdala
Resting Cerebral Blood Flow (CBF) | Baseline
  CBF derived from resting arterial spin labeled MRI
FMRI: Multisensory task activity | Baseline
  BOLD activation during multisensory task
FMRI: Spatial task activity | Baseline
  BOLD activation during spatial summation and divided attention
FMRI: BOLD resting connectivity of the posterior parietal cortex | Baseline
  BOLD resting connectivity of the posterior parietal cortex
FMRI: Graphesthesia Activation | Baseline
  BOLD activation during graphesthesia task
Pain Ratings | Baseline
  Visual analog scale (VAS) ratings of pain intensity and pain unpleasantness. The VAS is a scale of 0-10, with higher scores indicating a worse outcome.
Pain Ratings | 1 Year Followup
  Visual analog scale (VAS) ratings of pain intensity and pain unpleasantness. The VAS is a scale of 0-10, with higher scores indicating a worse outcome.
Spatial Distribution of Pain | Baseline
  Body map assessment of location of pain
Spatial Distribution of Pain | 1 Year Followup
  Body map assessment of location of pain

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coghill, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data That Will Be Shared:
  Data sharing represents a critical dimension of the proposed research. The data will be quite complex with psychological, psychophysical, demographic information collected outside of the scanner, and multiple modalities of MRI information collected during scanning. Accordingly, this rich dataset can be utilized for many secondary analyses. All modalities of data will be shared, with raw data included.
  Formatting of Data to Facilitate Sharing:
  As data is acquired, it will be named and placed into directory structures according to the BIDS standard (Brain Imaging Database Structure: http://bids.neuroimaging.io/). This standard accommodates all types of neuroimaging data to be acquired in the present proposal, and also allows for the inclusion of non-neuroimaging data such as psychological, psychophysical, and demographic information. Importantly, when data is in this format, it can be readily shared within OpenFMRI and other data warehouses
Supporting Information: SAP
Time Frame: Data will be made available after publication of key papers and will be permanently available with no expiration date.
Access Criteria: After publication of key papers, data will be freely available for all researchers.

DOCUMENTS (3):
  • Study Protocol (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05814497/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05814497/SAP_001.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT05814497/ICF_002.pdf